CLINICAL TRIAL: NCT05283018
Title: Continuous Monitoring of the P3a Response During General Anesthesia Using the Rough Auditory Stimuli Coupled to the Analysis of Frontal EEG Signal
Brief Title: Relationship Between the Depth of Anesthesia and Auditory Evoked Potentials (P3a)
Acronym: MP3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); Laboratoire de Mécanique des Solides, École polytechnique (Unknown); M3DISIM Inria Université Paris-Saclay (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP211287; 2021-A02322-39 (Other: IDRCB)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: General Anesthesia
Keywords: Auditory Evoked Potentials; Electroencephalography Phase Synchronization; P3 Event-Related Potentials; Depth of anesthesia; Acoustic Stimulation
MeSH Terms: interventions — Acoustic Stimulation; Ultrasonography, Doppler, Transcranial; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery under general anesthesia: Patients undergoing urgent or scheduled surgery at Lariboisière Hospital
  Interventions: Device: Electroencephalogram recording; Other: Auditory stimulation; Device: Transcranial Doppler; Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Electroencephalogram recording — Brain function monitoring using a Sedline® module (Masimo corporation) to evaluate the state of the brain under anesthesia
Other: Auditory stimulation — Monotonous sounds are sent via binaural headphones: a standard item and a distractor item (rough sound). Each stimulus lasts about 300 ms and they are separated by 1.5 to 2 seconds between them; the deviant sound/standard sound ratio is fixed between 1/5 and 1/6.
Device: Transcranial Doppler — Measurement of cerebral blood flow velocity (CFV) with use of Transcranial Doppler ultrasonography. For all patients, CFV (unit cm/s) will be collected over four distinct periods: 1/ baseline or during pre-oxygenation at inspired oxygen fraction (FiO2) of 21% in awake patients; 2/ during anesthetic induction; 3 /deep sleep; 4/ recovery period.
Device: Near-infrared spectroscopy — Continuous measurement of cerebral oxygen saturation (SO2) with Near-infrared spectroscopy (NIRS).
  For all patients, SO2 (%) will be collected over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3 /deep sleep; 4/ recovery period.

SUMMARY:
The interest of perioperative cerebral monitoring and in particular electroencephalography (EEG) to reduce neurological and cognitive damage in surgery has been the subject of abundant research and corresponds to a crucial issue. There is increasing evidence to suggest that inadequate (overdosed) anesthesia for patient characteristics and intraoperative hemodynamic instability is associated with an increased risk of complications including postoperative cognitive dysfunction and postoperative mortality.

However, these devices have many limitations in use, in particular their consideration of the muscle component of the electrical signal collected.There are other identifiable EEG signals that can be used to assess the depth of anesthesia, in particular auditory evoked potentials (AEPs).

The so-called rough sound waves correspond to a formulation composed of the rapid repetition of acoustic segments, at a frequency of 30 to 150 Hz.This frequency (whether sound or light) induces a temporal activation that captures attention and provokes unpleasant sensations and avoidance strategies when perceived by a subject.

This project aims at overcoming the interaction of the muscular electrical signal by evaluating the electrophysiological response (auditory evoked potentials) to particular sound stimuli, called "rough", thus underpinning the understanding of the mechanisms of neurosensory integration and attention during a state of loss of consciousness or altered consciousness.

The hypothesis proposed for this study is the following: the P3a wave (positive wave collected on the EEG during auditory evoked potentials) is altered during general anesthesia, in frequency and amplitude, and thus is indicative of the depth of the anesthetic state.

DETAILED DESCRIPTION:
Monitoring the depth of anesthesia remains a challenge for anesthesiologists. There is increasing evidence to suggest that inadequate (overdosed) anesthesia for patient characteristics and intraoperative hemodynamic instability is associated with an increased risk of postoperative complications and mortality.

Monitoring of cortical electroencephalogram (EEG) analysis has developed over time to address three daily issues:

* Prevention of hypnotic overdose
* The prevention of hypnotic underdosing, exposing to an increased risk of explicit perianesthetic memory
* The discussed relationship between a poor electroencephalographic trace, associated with a lowered blood pressure and a low dose of hypnotics used, and mortality at a distance from the anesthetic act (triple low concept).

However, these devices have many limitations in use, in particular their consideration of the muscle component of the electrical signal collected.

However, there are other identifiable EEG signals that can be used to assess the depth of anesthesia, in particular auditory evoked potentials.

The technique currently used to monitor the depth of anesthesia is the measurement of the bispectral index. However, this technique has its limits of use linked to the possible modifications of their interpretability by certain pharmacological agents (ketamine, high dose morphinics, Neuromuscular blockers, beta-blockers and ephedrine), by the electric scalpel and by persistent muscle contractions. In addition, the delay in analysis (about 30 seconds) may delay the interpretation of the result and the resulting therapeutic interventions.

The study of auditory evoked potentials seems to provide an alternative. Indeed, it has been shown in several studies that the P300 wave (or P3), a positive wave appearing at 300ms of stimulation) is partially inhibited by anesthesia and that its amplitude could be correlated to its depth.

These P300 waves are not affected by the different factors that can disturb the analysis of the bispectral index.

The rapid repetition of a sound or light signal produces a marked activation of certain neuronal chains in the temporal areas, particularly involved in the field of attention. This can induce undesired sensations and promote avoidance and distancing from the source. The repetition of a signal at a frequency of 40 to 80 Hz is perceived as particularly provoking.

Rough sounds synchronize auditory cortical regions as well as some frontal and limbic cortical regions and other subcortical regions.

This also suggests that the negative perception of rough sounds would be related to their ability to take control of neural networks usually involved in negative emotions and pain integration

The hypothesis proposed for this study is the following: the P3a wave (positive wave collected on the EEG during auditory evoked potentials) is altered during general anesthesia, in frequency and amplitude, and thus is indicative of the depth of the anesthetic state

Patients over 18 years old are eligible to participate in this protocol. During the anaesthesia consultation, they will be given a letter of information on the objectives and progress of the study. Their non-opposition to participating in this study will be collected at the latest during the pre-anaesthetic visit, the day before the operation, after a period of reflection. The patient will be offered to listen to the sounds used during this visit.

The protocol will start on the day of the operation. The procedures will be performed under general anesthesia. The protocol does not interact with the care procedure.

On the day of the procedure, a headset that is not a medical device is placed on the patient's ears. The P3a wave is collected using the EEG headband used in the operating room (Bispectral Index-BIS or PSI) to monitor the depth of anesthesia. The detection of this wave involves a post-processing phase of the signal and does not influence the anesthetist in charge of the patient.

The remaining non-invasive monitoring of brain function includes frontal EEG (Bispectral Index, BIS), bilateral transcranial Doppler, and a NIRS sensor used routinely for this type of procedure.

No invasive devices were used in addition to those required for anesthesia. All the monitoring instruments described above, except the one studied, are already used routinely in the department. The duration of anesthesia is not prolonged for the study.

The sound signals are emitted during the awake phase, the anesthetic induction and the awakening phase.

No additional examination will be performed. The anesthetic strategy is decided by the anesthesiologist in charge of the procedure.

The physician in charge of the study collecting the data does not intervene at any time in the management of the patient. The measures cannot influence the prescribing physician since at this stage the data are not yet analyzed and available.

Pilot study: No calculation of the number of subjects required due to the lack of comparable published data.

Effect size: In a reference article describing the effect of propofol during general anesthesia on P3 wave amplitude and latency, the observed variations in P3 wave latency were of the order of 50%.

Moreover, the proportion of patients for whom a sufficient depth of anesthesia is not reached with discordance between the bispectral index and the clinic is 20%. Assuming in the first group a latency μ_1=50% with a standard deviation of 10% and in the second group μ_1= 30% with a standard deviation of 20%. The sample size required to reject the H0 hypothesis: μ_1=μ_2 with a significance level of 0.05 and a power of 80% (1 - Type II error) via a Wilcoxon-Mann-Whitney test is N= 43 patients.

A target of 50 patients seems relevant.

The variations of P3 during induction and wake-up will be tested using a Student-t test after testing the normality of the distribution. The correlation between P3 variations and variations of EEG features (Burst suppression, SEF95) during induction and wake-up will be done using Pearson test. A full multivariate analysis will also be performed. All statistical analyses will be performed using R statistical software (The 'R' Foundation for Statistical Computing, Vienna, Austria). Results will be expressed as means (± standard deviation). A p-value of less than 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (≥ 18 years old)
* Eligible for an outpatient or scheduled surgery procedure under general anesthesia
* Patient who expressed his non-opposition to participation in this research

Exclusion Criteria:

* Patient under the age of 18
* Pre-existing auditory sensorineural impairment
* Severe pre-existing cognitive impairment (preoperative mini-mental state examination MMSE < 24)
* Patient opposed to participation in the protocol
* Pregnant woman
* Patient under judicial protection measure
* Patient without affiliation to a social security scheme
* Patient benefiting from the State medical assistance (AME) programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients eligible for an outpatient or scheduled surgery procedure under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Duration of the P3a subcomponent of the P300 | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  EEG monitoring of the P3a wave obtained by emission of rough sound signals: duration of P3a (ms) wave onset periods over four distinct periods: 1/baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
P3a amplitude | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  EEG monitoring of the P3a wave obtained by emission of rough sound signals: P3a amplitude (A in µV) over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
P3a frequency | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  EEG monitoring of the P3a wave obtained by emission of rough sound signals: P3a wave frequency (FP3 in Hz) over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
Depth of anesthesia | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  Depth of anesthesia measured by bispectral index (BIS, MASIMO, %) over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.

SECONDARY OUTCOMES:
Mean arterial blood pressure | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, the mean arterial pressure (mmHg) will be collected continuously, over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
Cerebral blood flow velocity (CFV) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, CFV (unit cm/s) will be collected continuously, using Transcranial Doppler, over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
Burst Suppression (BS) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, continuous measurement of BS duration (%) over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
Spectral Edge Frequency (SEF95) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, continuous measurement of SEF95 on intraoperative EEG - BIS in %, over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.
Cerebral oxygen saturation | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, the cerebral oxygen saturation (SO2; %) will be collected continuously using NIRS over four distinct periods: 1/ baseline or during pre-oxygenation at FiO2 of 21% in awake patients; 2/ during anesthetic induction; 3/ deep sleep; 4/ recovery period.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Fabrice VALLEE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care, Paris, France